CLINICAL TRIAL: NCT00663572
Title: Food Habit Programming: Influence of Genetics and Early Nutrition in a Population of Preterm Infants
Acronym: Polynuca
Status: Terminated | Type: Observational
Sponsor: Nantes University Hospital (Other)
Other Study IDs: BRD07/12-L; ID RCB 2007-A01432-51
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Preterm Infants
Keywords: Newborn; nutrition; genetic; feeding behaviour; psychomotor development; long-term effects; nutritional imprinting.
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Influence of neonatal nutrition and growth on psychomotor development of 2 years preterm infants.-Joint influence of environmental factor (early nutrition) and genetics factors on feeding behaviour setting- up in a particular population of infants of whom nutrition and life conditions during first weeks of life were purely controlled.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants < 33 SA who stayed at least 2 weeks after birth in Nantes hospital, included in the " Grandir ensemble " network, 2 years old in 2008 and 2009

Ages: 2 Years to 25 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants < 33 SA who stayed at least 2 weeks after birth in Nantes hospital, included in the " Grandir ensemble " network, 2 years old in 2008 and 2009
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental evaluation by ASQ (Age and stages Questionnaire) at 2 years of age | 2 years of age

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Nantes, Nantes, France

REFERENCES:
- [Derived] Migraine A, Nicklaus S, Parnet P, Lange C, Monnery-Patris S, Des Robert C, Darmaun D, Flamant C, Amarger V, Roze JC. Effect of preterm birth and birth weight on eating behavior at 2 y of age. Am J Clin Nutr. 2013 Jun;97(6):1270-7. doi: 10.3945/ajcn.112.051151. Epub 2013 Apr 24. PMID 23615831